CLINICAL TRIAL: NCT01290250
Title: Evaluation of a New Orange-Based Beverage Enriched With Polyphenols (Whole Press) on Features of Metabolic Syndrome and Cardiovascular Risk Factors Related to Inflammation and Antioxidant Defense System in Adult Humans
Brief Title: Evaluation of a New Orange-Based Beverage Enriched With Polyphenols in Adult Humans
Acronym: BIONAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Coca-Cola Company (Industry)
Responsible Party: Principal Investigator, Concepcion Aguilera, Lecturer of Biochemistry and Molecular Biology, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BIONAOS-ORANGE
Record Dates: First submitted 2010-12-21; First posted 2011-02-04 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orange juice based beverage enriched in polyphenols (Experimental): 2 daily doses (250 ml each) during 3 months
  Interventions: Other: Orange juice based beverage enriched in polyphenols
- Orange juice with low levels of polyphenols (Placebo Comparator): 2 daily doses (250 ml each) during 3 months
  Interventions: Other: Orange juice based beverage enriched in polyphenols

INTERVENTIONS:
Other: Orange juice based beverage enriched in polyphenols — 2 daily doses (250 ml each) during 3 months

SUMMARY:
The purpose of this study is to evaluate the effects of a new orange juice-based beverage enriched in fiber and selected phenolic compounds (mainly flavanones) on features of metabolic syndrome and cardiovascular disease risk factors related to inflammation and antioxidant defense system in overweight and obese adult humans. This study hypothesizes that consumption of an orange juice-based beverage enriched in fiber and selected phenolic compounds (mainly flavanones)would improve lipid levels and lipid metabolism,blood pressure and the Homeostatic Model Assessment (HOMA) index.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) higher than 25 (overweight or obese) but lower than 40 (extreme obesity) or waist circumference higher than 94 cm for men and 80 cm for women,

and having altered at least two markers of MS namely:

* Hypertension (diastolic pressure higher than 85 mmHg but lower than 110 mmHg)
* Hyperglycemia (higher than 100 mg/dl but lower than 130 mg/dl)
* Elevated plasma triacylglycerol concentrations (higher than 150 mg/dl)
* Decreased plasma HDL-c levels (lower than 40 for men and 50 for women)
* Volunteers will be otherwise healthy and without taking any medication aiming to lower either blood lipids, blood pressure or blood glucose concentrations.

Exclusion Criteria:

* The presence of morbid obesity
* Blood pressure higher than 110 mmHg
* Plasma glucose levels higher than 130 mg/dl
* The use of any medication for the control of blood pressure or glucose or lipid metabolism
* Medical history of consumption of hypocaloric diet in the last year
* Disorders of the food conduct
* The presence of familiar dislipemias relatives of genetic character or the denial to take part in the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 months
Fasting Plasma Insulin Concentration | 3 months
Fasting Plasma Triacylglycerols Concentration | 3 months
Fasting Plasma High-Density Lipoprotein Cholesterol Concentration | 3 months
Insulin resistance using HOMA (Homeostatic Model Assessment)index | 3 months
  The HOMA index will be calculated as the product of the fasting plasma insulin level (mU/mL) and the fasting plasma glucose level (mmol/L), divided by 22.5
Fasting Plasma glucose concentrations | 3 months
Diastolic blood pressure | 3 months

SECONDARY OUTCOMES:
Antioxidant defense system | 3 months
  Biomarkers of the non-enzymatic (NE-ADS) and enzymatic antioxidant defense system (E-ADS). For the NE-ADS, in addition to total plasma antioxidant capacity, malondialdhyde, and total carbonyl protein derivatives, plasma α-tocopherol, β-carotene, retinol, coenzyme Q and total blood glutathione will be determined. Furthermore, the amount of plasma oxidized LDL and urinary 8-hydroxy-2'-deoxyguanosine and F2-isoprostanes will be measured. For E-ADS the activities of glutathione reductase, glutathione peroxidase, superoxide dismutase, and catalase in red blood cells will be assessed.
Biomarkers of inflammation | 3 months
  Biomarkers of inflammation: Interleukin-1 beta (IL-1β), interleukin-6 (IL-6), interleukin-8 (IL-8), matrix metalloproteinase-9 (MMP-9), monocyte chemotactic protein 1 (MCP-1)and polymorphonuclear neutrophils myeloperoxidase (MPO)
Biomarkers of cardiovascular risk. | 3 months
  Biomarkers of cardiovascular risk:soluble endothelial selectin (sE-selectin), soluble intercellular adhesion molecule 1 (sICAM-1), soluble vascular cell adhesion molecule (sVCAM-1), total and active tissue plasminogen activator inhibitor-1 (tPAI-1), tumor necrosis factor alpha (TNF-α).
Metabolic analysis | 3 months
  Gastrointestinal hormones involved in the control of satiety and insulin secretion i.e. active amylin, ghrelin (GHR), glucagon peptide-1 (GLP-1), gastric inhibitory peptide or gastric insulinotropic peptide (GIP), polypeptide YY 3-36, pancreatic polypeptide (PP).
  Likewise, adiponectin, leptin, resistin, visfatin, hepatocyte growth factor (HGF), nerve growth factor (NGF), retinol binding protein 4 (RBP4) and L-fatty acid binding protein (L-FABP) will be determined
Gene expression analysis | 3 months
  Whole genome gene expression analysis: This analysis will be carried out in a subset of 20 control and 20 experimental samples at four times: 160 arrays. The GeneChip® Human Exon 1.0 ST will be used for the gene expression analysis.
  Validation by Reverse transcription polymerase chain reaction (RTPCR): In order to confirm the arrays results, a total of 93 differentially expressed genes in the experimental samples will be analyzed by RTPCR using low density arrays

CONTACTS AND LOCATIONS:
Overall Officials: Concepcion Aguilera, Phd, Principal Investigator — Universidad de Granada; Maria Dolores Mesa, PhD, Principal Investigator — Universidad de Granada; Angel Gil, PhD, Study Chair — Universidad de Granada
Locations (1):
- Department of Biochemistry and Molecular Biology II, Institute of Nutrition and Food Technology, Center for Biomedical Research, University of, Granada, Granada, Spain

REFERENCES:
- [Derived] Rangel-Huerta OD, Aguilera CM, Martin MV, Soto MJ, Rico MC, Vallejo F, Tomas-Barberan F, Perez-de-la-Cruz AJ, Gil A, Mesa MD. Normal or High Polyphenol Concentration in Orange Juice Affects Antioxidant Activity, Blood Pressure, and Body Weight in Obese or Overweight Adults. J Nutr. 2015 Aug;145(8):1808-16. doi: 10.3945/jn.115.213660. Epub 2015 Jul 1. PMID 26136593